CLINICAL TRIAL: NCT06872034
Title: The Efficacy and Safety of Venostan (Horse Chestnut Seed Extract Tablets) in Promoting Postoperative Swelling Reduction in Patients With Ankle Fractures: A Multicenter, Open-Label, Randomized Controlled Trial
Brief Title: The Efficacy and Safety of Venostan in Promoting Postoperative Swelling Reduction in Patients With Ankle Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, LiTing, Chief Physician, Beijing Jishuitan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K2025-003-00
Record Dates: First submitted 2025-02-27; First posted 2025-03-12 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-04

CONDITIONS: Swelling/ Edema
Keywords: Ankle fracture; Edema; Postoperative rehabilitation; horse chestnut seed extract; venostan; enhanced recovery after surgery
MeSH Terms: conditions — Edema; Ankle Fractures | interventions — venostasin; horse chestnut seed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Venostan (horse chestnut seed extract tablets) (Experimental)
  Interventions: Drug: Venostasin (horse chestnut seed extract tablets); Other: standard treatment
- control (Other)
  Interventions: Other: standard treatment

INTERVENTIONS:
Drug: Venostasin (horse chestnut seed extract tablets) — Venostasin (horse chestnut seed extract tablets) ，twice daily, 400 mg per dose, for 14 days
  Arms: Venostan (horse chestnut seed extract tablets)
Other: standard treatment — standard treatment

SUMMARY:
This study is a multicenter, open-label, randomized controlled trial planned to enroll patients with ankle fractures who meet the inclusion and exclusion criteria and are scheduled to undergo internal fixation surgery from the emergency and inpatient wards of multiple hospitals. General and disease-related data will be collected. All eligible patients must voluntarily sign an informed consent form after understanding and accepting the study. Successfully recruited participants will undergo internal fixation surgery at a scheduled time and then be randomly assigned to either the Venostan (horse chestnut seed extract tablet) group or the conventional treatment group. They will receive the corresponding treatments according to the study protocol. Follow-up assessments will include changes in ankle circumference, ankle range of motion, scale evaluation results, laboratory test results, and adverse events. The study aims to evaluate the effects of Venostasin in patients with ankle fractures undergoing internal fixation surgery, exploring its potential to promote postoperative reduction of ankle swelling, enhance early joint function recovery, and investigate its safety in postoperative fracture management.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 year old, no gender restriction;
* Diagnosed with ankle fracture confirmed by imaging data, AO classification: ---AO-43, AO-44-F3, AO-44;
* Scheduled to undergo open reduction and internal fixation surgery;
* Voluntary signing of the informed consent form.

Exclusion Criteria:

* Pregnant or lactating women;
* With contraindications to surgery;
* With other severe combined injuries or soft tissue infections;
* Severe multiple trauma: Injury Severity Score (ISS) > 16;
* With concurrent fractures of the spine, pelvis, or ipsilateral or contralateral lower limbs;
* Pathological fractures;
* With peripheral vascular disease or deep vein thrombosis (DVT);
* With severe impairment of heart, lung, liver, or kidney function or abnormal coagulation function;
* Unable to walk independently before the injury;
* With pre-existing lower limb edema (e.g., due to liver cirrhosis, kidney disease, etc.) before the injury;
* With mental disorders or hyperalgesia;
* Allergic to any component of the investigational drug;
* Any contraindications that limit clinical evaluation and treatment of the patient;
* Deemed unsuitable for inclusion in this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-01-12 (Estimated); Study Completion 2026-01-12 (Estimated)

PRIMARY OUTCOMES:
Change in ankle circumference at 6 days postoperatively compared to baseline | from enrollment to the 6th day postoperation
  Defined as the change in ankle circumference measured using the figure-of-eight method on postoperative day 6 (after 5 days of Venostan treatment) compared to the ankle circumference measured on postoperative day 2 (before the first dose of Venostan)

SECONDARY OUTCOMES:
Change in ankle circumference at 14 days postoperatively compared to baseline | from enrollment to the 14th day postoperation
  Defined as the change in ankle circumference measured using the figure-of-eight method on postoperative day 14 (after 13 days of Venostan treatment) compared to the ankle circumference measured on postoperative day 2 (before the first dose of Venostan)
Percentage change in ankle circumference at 6 and 14 days postoperatively compared to baseline | from enrollment to the 14th day postoperation
  Defined as the percentage change in ankle circumference measured using the figure-of-eight method on postoperative days 6 and 14 (after 5 and 13 days of Venostan treatment, respectively) compared to the ankle circumference measured on postoperative day 2 (before the first dose of Venostan)
Change in Visual Analog Scale (VAS) pain score at 6 and 14 days postoperatively | from enrollment to the 14th day postoperation
  Defined as the change in the patient-reported Visual Analog Scale (VAS) pain score on postoperative days 6 and 14 (after 5 and 13 days of Venostan treatment, respectively) compared to the score on postoperative day 2，VAS range from 0 to 10, and higher scores mean a worse outcome
EuroQol-5 dimension (EQ-5D) score at 6 and 14 days postoperatively | from enrollment to the 14th day postoperation
  Defined as the EuroQol-5 dimension (EQ-5D) quality of life score reported by the patient on postoperative days 6 and 14 (after 5 and 13 days of Venostan treatment, respectively), EQ-5D consists of 5 dimension, and every dimension consists of 5 level, the higher lever means a worse outcome
Ankle range of motion at 6 and 14 days postoperatively | from enrollment to the 14th day postoperation
  Defined as the ankle range of motion assessed by the investigator through physical examination on postoperative days 6 and 14 (after 5 and 13 days of Venostan treatment, respectively)
Incidence of deep vein thrombosis (DVT) in the lower limbs within 14 days postoperatively | from enrollment to the 14th day postoperation
  Defined as the incidence of deep vein thrombosis (DVT) detected by lower limb vascular ultrasound within 14 days postoperatively
Rate of surgical complications | from enrollment to 30 days after discontinuation of medication
  Defined as complications related to the fracture surgery, with the severity of complications assessed by the investigator using the Clavien-Dindo classification of surgical complications

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Jishuitan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No